CLINICAL TRIAL: NCT01673048
Title: From Bench to Bedside: Modification of Elastic Stable Intramedullary Nailing With a 3rd Nail in a Femoral Spiral Fracture Model and Its Transmission to Clinical Practice
Brief Title: Modification of ESIN-osteosynthesis in a Femoral Fracture Model and Its Transmission to Clinical Practice
Acronym: ESIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Martin M Kaiser, Consultant, University of Luebeck
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3ESINFemur
Record Dates: First submitted 2012-08-12; First posted 2012-08-27 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Femoral Fracture; Children
Keywords: Elastic stable intramedullary nailing; biomechanical testing; fracture; femur; treatment; children; adolescents
MeSH Terms: conditions — Femoral Fractures; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Femoral fracture, ESIN (Active Comparator): Prospectively all patients treated with the 3-nail-configuration for dislocated femoral shaft fractures were enrolled; 25 patients are planned, 18 could be enrolled Comparison will be with own previous data of patients treated with the "classical" 2-C-shaped ESIN-osteosynthesis
  Interventions: Procedure: 3-Nail-ESIN in femoral shaft fractures

INTERVENTIONS:
Procedure: 3-Nail-ESIN in femoral shaft fractures

SUMMARY:
Elastic stable intramedullary nailing (ESIN) is the standard treatment for displaced diaphyseal femoral fractures in children. However, some literature report high complication rates (10-50%) in complex fractures. Data of our own patients with special emphasis on complications showed also mediocre results. Thus, a biomechanical study was conducted to search for modifications. In this study the stiffness with a 3rd nail implanted was compared to the classical 2 C-shaped configuration. For each of the 3 configurations of retrograde ESIN (titanium nails) eight composite femoral grafts (Sawbones®) with an identical spiral fracture were used: 2C configuration (2 C-shaped nails, 2x3.5 mm), 3CM configuration (3rd from antero-medial, + 1x2.5 mm) and 3CL configuration (3rd from antero-lateral, + 1x2.5 mm). Each group underwent biomechanical testing in 4-point bending, IRO/ERO and axial compression (0°/9°). Due to a significantly higher stiffness of 3CL in the anterior-posterior, internal rotation and 9° compression directions implantation of 3 nails became standard treatment for all dislocated femoral fractures at our department.

All patients were followed prospectively. The following data was collected: Type of osteosynthesis, any kind of complication (additional procedures like cast or external fixateur, Re-Do operations, misalignment, pseudarthrosis, skin irritation, infection), time until full weight bearing and time until implant removal. At follow-up the legs were controlled for a possible length discrepancy and a possible deviation of axis. Patients' satisfaction was controlled by CSQ (clients satisfaction score, Larsen et al 2002). Further on the Harris Hip Score was used. X-ray controls were done as standard care protocol after 1 and 3-4 months (dependend on age).

Level of Evidence IV Keywords: Elastic stable intramedullary nailing, biomechanical testing, fracture, femur, treatment, children, adolescents.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Dislocated femoral fracture
* ESIN osteosynthesis

Exclusion Criteria:

* No given informed consent
* Other osteosynthesis than ESIN

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2009-01; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Intraoperative and postoperative complications | 12 months
  All complications will be recorded: Intraoperative and postoperative complications, Re-Do operations

SECONDARY OUTCOMES:
misalignment | 12 m
  Follow up X-rays will be measured for misalignment in degrees (sagittal, frontal and transverse plane) Data will be grouped as
  a) 1 - 5° b) 6 - 10° c) 11 - 15° d)16 - 20° e) 20 - 30° f) > 30°
Pseudarthrosis | 12 m

OTHER OUTCOMES:
Limb discrepancy | 12 m
  both legs will be measured from spina iliaca anterior superior to the lateral malleolus in cm.
  Results will be grouped as:
  a) 0 - 0.5 cm b) 0.6 - 1.0 cm c) 1.1 - 1.5 cm d) 1.6 - 2.0 cm e)> 2 cm

CONTACTS AND LOCATIONS:
Overall Officials: Martin M Kaiser, PD Dr. med., Principal Investigator — University Luebeck
Locations (1):
- Department of Pediatric Surgery, Lübeck, Germany

REFERENCES:
- [Background] Kaiser MM, Zachert G, Wendlandt R, Eggert R, Stratmann C, Gros N, Schulze-Hessing M, Rapp M. Increasing stability by pre-bending the nails in elastic stable intramedullary nailing: a biomechanical analysis of a synthetic femoral spiral fracture model. J Bone Joint Surg Br. 2012 May;94(5):713-8. doi: 10.1302/0301-620X.94B5.28247. PMID 22529097
- [Background] Kaiser MM, Zachert G, Wendlandt R, Rapp M, Eggert R, Stratmann C, Wessel LM, Schulz AP, Kienast BJ. Biomechanical analysis of a synthetic femoral spiral fracture model: Do end caps improve retrograde flexible intramedullary nail fixation? J Orthop Surg Res. 2011 Sep 18;6:46. doi: 10.1186/1749-799X-6-46. PMID 21923948
- [Background] Kaiser MM, Wessel LM, Zachert G, Stratmann C, Eggert R, Gros N, Schulze-Hessing M, Kienast B, Rapp M. Biomechanical analysis of a synthetic femur spiral fracture model: Influence of different materials on the stiffness in flexible intramedullary nailing. Clin Biomech (Bristol). 2011 Jul;26(6):592-7. doi: 10.1016/j.clinbiomech.2011.01.012. Epub 2011 Feb 22. PMID 21345557
- [Result] Kaiser MM, Stratmann C, Zachert G, Schulze-Hessing M, Gros N, Eggert R, Rapp M. Modification of elastic stable intramedullary nailing with a 3rd nail in a femoral spiral fracture model - results of biomechanical testing and a prospective clinical study. BMC Musculoskelet Disord. 2014 Jan 8;15:3. doi: 10.1186/1471-2474-15-3. PMID 24397612
- See also: Department of Pediatric Surgery Luebeck — http://www.kinderchirurgie.uni-luebeck.de/